CLINICAL TRIAL: NCT06264063
Title: Study of Behavioral Dysfunctions and Related Neuronal Correlates in Patients With Dystonia
Acronym: D-DIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Caterina Formica, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: D-DIST
Record Dates: First submitted 2023-12-28; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: Dystonia; Neurologic Disorder; NEUROSCIENCE
MeSH Terms: conditions — Dystonia; Nervous System Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): patients with dystonia were submitted to a neuropsychological evaluation
  Interventions: Behavioral: experimental group; Diagnostic Test: EEG power in alpha band
- control group (Experimental): healthy patients were submitted to a neuropsychological evaluation
  Interventions: Behavioral: control group; Diagnostic Test: EEG power in alpha band

INTERVENTIONS:
Behavioral: control group — the investigators have to assess the neuropsychological and psychological profile with specific questionnaire that evaluated the moral index, presence of obsessive and compulsive disorders and Montreal Cognitive Assessment to evaluate cognitive functions
  Arms: control group
Behavioral: experimental group — the investigators have to assess the neuropsychological and psychological profile with specific questionnaire that evaluated the moral index, presence of obsessive and compulsive disorders and Montreal Cognitive Assessment to evaluate cognitive functions
  Arms: experimental group
Diagnostic Test: EEG power in alpha band — partecipants were submitted to registration of electrical activity with EEG to study the EEG power in alpha band

SUMMARY:
Dystonias represent hyperkinetic movement disorders characterized by protracted muscle contractions, such as to cause torsional movements and anomalous postures in different parts of the body. Although they occur more often in a focal form (blepharospasm, oromandibular dystonia, cervical dystonia, laryngeal dystonia, attitudinal cramps of the limbs) than segmental (involvement of several contiguous muscle groups, e.g. facial muscles and neck muscles), they are nevertheless capable of significantly influencing the quality of life, with consequent social and health costs. Although described as a predominantly motor disorder, the presence of non-motor symptoms in dystonias associated with alteration of the fronto-striatal circuits is increasingly recognized. Neuroimaging studies have highlighted that the striatum and, more specifically, striatal dopamine, is involved in high cognitive processes such as attention, reward-based learning and decision making. Clinical conditions associated with cortico-striatal circuit dysfunction and abnormal meso-striatal or meso-cortical dopamine transmission also appear to influence temporal estimation, delay discounting, showing an impulsive preference for immediate rewards over delayed gratification.

Based on these premises, the present project aims to evaluate the cognitive and affective aspects of dystonias, in line with neuroimaging research documenting structural and functional dysfunctions in the respective brain regions.

DETAILED DESCRIPTION:
Dystonias represent hyperkinetic movement disorders characterized by protracted muscle contractions, such as to cause torsional movements and anomalous postures in different parts of the body. Although they occur more often in a focal form (blepharospasm, oromandibular dystonia, cervical dystonia, laryngeal dystonia, attitudinal cramps of the limbs) than segmental (involvement of several contiguous muscle groups, e.g. facial muscles and neck muscles), they are nevertheless capable of significantly influencing the quality of life, with consequent social and health costs. Although described as a predominantly motor disorder, the presence of non-motor symptoms in dystonias associated with alteration of the fronto-striatal circuits is increasingly recognized. Neuroimaging studies have highlighted that the striatum and, more specifically, striatal dopamine, is involved in high cognitive processes such as attention, reward-based learning and decision making. Clinical conditions associated with cortico-striatal circuit dysfunction and abnormal meso-striatal or meso-cortical dopamine transmission also appear to influence temporal estimation, delay discounting, showing an impulsive preference for immediate rewards over delayed gratification.

Based on these premises, the present project aims to evaluate the cognitive and affective aspects of dystonias, in line with neuroimaging research documenting structural and functional dysfunctions in the respective brain regions.

The study aims to investigate the neurocognitive profile in patients with dystonia. In particular, investigators will evaluate the correlation between the alterations of the subcortical areas and the cognitive and affective functions involved in the processes of evaluating risk, reward and impulsivity.

Primary Objectives:

Study of cognitive and affective functions in dystonic subjects, with particular reference to the mechanisms of reward learning, inhibitory control and impulsivity.

Secondary objectives:

Connectivity analysis of neuronal substrates related to higher order cognitive alterations

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old;
* Informed consent;
* Montreal cognitive assessment > 21;

Exclusion Criteria:

* Patients with cervical dystonia with anterocollis spasm;
* Sensory-motor deficits that can hinder neuropsychological assessment
* Contraindications to performing Magnetic Resonance Imaging

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
montreal cognitive assessment | 1 hour
  Study of cognitive functions in dystonic subjects, with particular reference to the mechanisms of memory, attention and executive functions
Beck depression inventory | 1 hour
  Study of affective functions in dystonic subjects, with particular reference to the mechanisms of mood and evaluating the presence of depressive symptoms

SECONDARY OUTCOMES:
EEG power in alpha band | 1 hour
  Connectivity analysis of neuronal substrates related to higher order cognitive alterations and the power of alpha band

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy